CLINICAL TRIAL: NCT05596474
Title: Application of Beet-root Juice Supplementation and Photobiomodulation Treatment on Forearm Muscle Fatigue in Older Adults
Brief Title: Effect of Beet-root Juice and PBM Treatments on Muscle Fatigue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Principal Investigator, Andrew Wells, Ph.D, Principal Investigator, Wake Forest University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB00024675
Record Dates: First submitted 2022-10-21; First posted 2022-10-27 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Health Care Utilization; Healthy Aging
Keywords: Red light therapy; Forearm muscle endurance; Beet-root juice; Electromyography
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Beet-root juice plus red-light therapy (Experimental)
  Interventions: Dietary Supplement: Beet-root juice; Radiation: red-light therapy
- Beet-root juice plus sham light therapy (Sham Comparator)
  Interventions: Dietary Supplement: Beet-root juice; Radiation: sham light
- Placebo plus red-light therapy (Placebo Comparator)
  Interventions: Radiation: red-light therapy; Dietary Supplement: Placebo
- Placebo plus sham light therapy (Active Comparator)
  Interventions: Dietary Supplement: Placebo; Radiation: sham light

INTERVENTIONS:
Dietary Supplement: Beet-root juice — Two days prior to the forearm endurance protocol, participants will be provided and instructed to consume a 400mg nitrate once per day. On the day of the forearm endurance protocol, the participants will be provided and instructed to consume a third 400mg dose of nitrates at least 150 minutes before forearm endurance testing.
  Other Names: Beet it Sport
  Arms: Beet-root juice plus red-light therapy; Beet-root juice plus sham light therapy
Radiation: red-light therapy — Participants will place their dominant forearm 15 centimeters away from the light source and have their dominant forearm exposed to 660nm wave length light for 10-minutes.
  Other Names: MitoMIN
  Arms: Beet-root juice plus red-light therapy; Placebo plus red-light therapy
Dietary Supplement: Placebo — Two days prior to the forearm endurance protocol, participants will be provided and instructed to consume a nitrate depleted placebo once per day. On the day of the forearm endurance protocol, the participants will be provided and instructed to consume a third dose of the nitrate depleted placebo at least 150 minutes before forearm endurance testing.
  Arms: Placebo plus red-light therapy; Placebo plus sham light therapy
Radiation: sham light — Participants will place their dominant forearm 15 centimeters away from the light source and have their dominant forearm exposed to sham light for 10-minutes.
  Arms: Beet-root juice plus sham light therapy; Placebo plus sham light therapy

SUMMARY:
The goal of this randomized counterbalanced repeated measures study is to test beet-root juice supplementation and red light therapy augment forearm muscle endurance in apparently healthy older adults over 65 years of age. The main questions seek to answer the following question:

Does beet-root juice supplementation improve forearm muscle endurance compared to a placebo supplement?

Does red light therapy improve forearm muscle endurance compared to a sham light exposure?

Does beet-root juice supplementation in combination with red light therapy improve forearm muscle endurance compared to a placebo-sham light control?

ELIGIBILITY:
Inclusion Criteria:

* Self-reports performing at least 30 minutes of light to moderate intensity physical activity 3 times per week for the last three months

Exclusion Criteria:

* Currently smoke
* Have smoked within the last 6 months
* Are taking taking supplements known to increase blood nitrate levels
* Have a known kidney disease
* Have a known liver disease
* Have a known thyroid condition
* Have a known gastritis condition
* Are taking medications that are known to cause complications with nitrate supplementation
* Have known or reported joint pain within the dominant hand

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Total forearm work performed | During the forearm exercise fatigue protocol lasting up to 45 minutes
  Work is the product of the number of times the forearm is activated multiplied by the amount of force produced by the forearm in kilograms.

SECONDARY OUTCOMES:
Forearm endurance | During the forearm exercise fatigue protocol lasting up to 45 minutes
  The duration of time the participant takes to complete the forearm fatigue protocol
Intermuscular coordination | During the forearm exercise fatigue protocol lasting up to 45 minutes
  Surface electromyography measurements of muscle activity

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Wells, Ph.D., Principal Investigator — Wake Forest University, Reynolda Campus
Locations (1):
- Wake Forest Univesity, Winston-Salem, North Carolina, United States